CLINICAL TRIAL: NCT01433406
Title: Long-term Study of TAK-875
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Model: Parallel
Other Study IDs: TAK-875/OCT-002; U1111-1124-1561 (Registry Identifier: WHO); JapicCTI-111602 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2011-09-12; First posted 2011-09-14 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Diabetes Mellitus
Keywords: Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus | interventions — TAK-875

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAK-875 25 mg (Experimental): (long-term monotherapy or long-term combination therapy with anti-diabetic drugs)
  Interventions: Drug: TAK-875
- TAK-875 50 mg (Experimental): (long-term monotherapy or long-term combination therapy with anti-diabetic drugs)
  Interventions: Drug: TAK-875

INTERVENTIONS:
Drug: TAK-875
  Arms: TAK-875 25 mg
Drug: TAK-875
  Arms: TAK-875 50 mg

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of long-term treatment with TAK-875 in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is an outpatient.
2. The participant signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.

Exclusion Criteria:

1. The participant has any serious cardiac disease, serious cerebrovascular disorder, or any serious pancreatic or hematological disease.
2. The participant is considered ineligible for the study for any other reason by the investigator or sub-investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1222 (Actual)
Dates: Start 2011-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Adverse events | From Baseline to Week 53
  Frequency, severity, and time to onset of adverse drug reactions tabulated by each symptom. Adverse events are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug.

CONTACTS AND LOCATIONS:
Locations (71):
- Japan (71):
  - Nagoya, Aichi-ken
  - Chiba, Chiba
  - Funabashi-shi, Chiba
  - Katori-shi, Chiba
  - Kisarazu-shi, Chiba
  - Matsudo-shi, Chiba
  - Matsuyama, Ehime
  - Nihama-shi, Ehime
  - Saijo-shi, Ehime
  - Fukuoka, Fukuoka
  - Kitakyushu-shi, Fukuoka
  - Onga-gun, Fukuoka
  - Annaka-shi, Gunma
  - Takasaki-shi, Gunma
  - Aki-gun, Hiroshima
  - Hiroshima, Hiroshima
  - Chitose-shi, Hokkaido
  - Sapporo, Hokkaido
  - Amagasaki-shi, Hyōgo
  - Nishinomiya-shi, Hyōgo
  - Mito, Ibaragi
  - Naka, Ibaragi
  - Tsuchiura-shi, Ibaragi
  - Ushiku-shi, Ibaragi
  - Sakade-shi, Kagawa-ken
  - Izumi-shi, Kagoshima-ken
  - Kamakura-shi, Kanagawa
  - Yamato-shi, Kanagawa
  - Kochi, Kochi
  - Suzaki-shi, Kochi
  - Kumamoto, Kumamoto
  - Minamata-shi, Kumamoto
  - Uji-shi, Kyoto
  - Miyazaki, Miyazaki
  - Matsumoto-shi, Nagano
  - Nagasaki, Nagasaki
  - Omura-shi, Nagasaki
  - Ōita, Oita Prefecture
  - Okayama, Okayama-ken
  - Izumisano, Osaka
  - Kashiwara-shi, Osaka
  - Osaka, Osaka
  - Sakai-shi, Osaka
  - Suita-shi, Osaka
  - Toyonaka-shi, Osaka
  - Saga, Saga-ken
  - Fujimi-shi, Saitama
  - Saitama-shi, Saitama
  - Sayama-shi, Saitama
  - Tokorozawa-shi, Saitama
  - Ōtsu, Shiga
  - Fujinomiya-shi, Shizuoka
  - Shizuoka, Shizuoka
  - Shimotsuga-gun, Tochigi
  - Shimotsuke-shi, Tochigi
  - Komatsu-shi, Tokushima
  - Bunkyo-ku, Tokyo
  - Chiyoda-ku, Tokyo
  - Chuo-ku, Tokyo
  - Hino-shi, Tokyo
  - Itabashi-ku, Tokyo
  - Katsushika-ku, Tokyo
  - Mitaka-shi, Tokyo
  - Nerima-ku, Tokyo
  - Ōta-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Sibuya-ku, Tokyo
  - Toyoshima-ku, Tokyo
  - Sanyoonoda-shi, Yamaguchi
  - Shimonoseki-shi, Yamaguchi
  - Ube-shi, Yamaguchi